CLINICAL TRIAL: NCT03464487
Title: Comparison Between Efficacy of Daily and Intermittent Low Glycemic Index Therapy Diet Among Children With Drug Resistant Epilepsy Aged 1-15 Years: an Open Labeled Randomized Controlled Parallel Design Non-inferiority Trial
Brief Title: Comparison Between Efficacy of Daily and Intermittent Low Glycemic Index Therapy Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor and Chief, Child Neurology Division, Department of Pediatrics, AIIMS, New Delhi, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Daily vs Intermittent LGIT
Record Dates: First submitted 2018-01-01; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Drug Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily LGIT (Active Comparator): The children with drug resistant epilepsy in this arm will receive Low Glycemic Index Therapy diet everyday along with the antiepileptic drugs.
  Interventions: Dietary Supplement: Low Glycemic Index Therapy Diet
- Intermittent LGIT (Active Comparator): The children with drug resistant epilepsy in this arm will receive Low Glycemic Index Therapy Diet on five days of each week along with antiepileptic drugs. Rest of the two days, they will receive a liberal diet.
  Interventions: Dietary Supplement: Low Glycemic Index Therapy Diet

INTERVENTIONS:
Dietary Supplement: Low Glycemic Index Therapy Diet — Low Glycemic Index Therapy Diet allows only carbohydrates with Glycemic Index less than 50 and also restricts daily carbohydrate intake to less than 40-60 gram per day.

SUMMARY:
Drug resistant epilepsy constitutes about one third of all children diagnosed with epilepsy. Although ketogenic diet is being used for drug resistant epilepsy for almost hundred years, its restrictiveness and adverse effects interferes with its compliance. So less restrictive alternatives like Low Glycemic Index Therapy diet is gradually becoming more popular and its effectiveness is well established. Still the restrictiveness of such monotonous diets is one of the most significant issues for long term maintenance of children on dietary therapy. In this study, we are planning to compare the efficacy of daily and intermittent Low Glycemic Index therapy Diet in children aged 1-15 years with drug resistant epilepsy in a open labelled randomized controlled non-inferiority trial. The children in intermittent LGIT arm will receive the dietary therapy for five days of each week, alternating with a liberal diet on the rest of the two days of the week.

DETAILED DESCRIPTION:
Drug resistant epilepsy constitutes about one third of all children diagnosed with epilepsy. Although ketogenic diet is being used for drug resistant epilepsy for almost hundred years, its restrictiveness and adverse effects interferes with its compliance. So less restrictive alternatives like Low Glycemic Index Therapy diet is gradually becoming more popular and its effectiveness is well established. Still the restrictiveness of such monotonous diets is one of the most significant issues for long term maintenance of children on dietary therapy. In this study, we are planning to compare the efficacy of daily and intermittent Low Glycemic Index therapy Diet in children aged 1-15 years with drug resistant epilepsy in a open labelled randomized controlled non-inferiority trial. The children in intermittent LGIT arm will receive the dietary therapy for five days of each week, alternating with a liberal diet on the rest of the two days of the week. With a follow up period of 6 months, we are planning to enroll 55 children in each arm. Adverse effect profile in each arm will also be monitored during the study. Also the effect of the dietary therapy on behavior and cognition in each arm will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 1-15 years with drug resistant epilepsy
2. Willing to come for regular follow up

Exclusion Criteria:

1. Surgically remediable cause for drug resistant epilepsy
2. Proven in born error of metabolism except in which dietary therapy for epilepsy is indicated(i.e. pyruvate carboxylase deficiency and GLUT 1 deficiency)
3. Previously received KD, MAD or LGIT
4. Known case of

   * Chronic kidney disease
   * Chronic liver disease/GI illness
   * Chronic heart disease(congenital and acquired)
   * Chronic respiratory illness

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of seizure reduction from baseline at 24 weeks in each arm | Percentage seizure reduction will be calculated for each child in each arm after 24 weeks follow up period is completed and finally mean seizure reduction in each arm will be computed at the end of 24 weeks
  Percentage of seizure reduction from baseline at 24 weeks in each arm will be calculated from Daily Seizure Log maintained by parents Percentage of seizure reduction at 24 weeks=x-y/x X 100 Y=Mean daily seizures at 24 weeks as measured over past 4 weeks X=Mean daily seizures at baseline as measured over 4 weeks Seizure log will contain details of number, duration and type of seizures as recorded by parents

SECONDARY OUTCOMES:
Proportion of patients with >50% seizure reduction in each dietary arm | At the end of 24 weeks, it will be determined the proportion of children in each arm with >50% reduction in seizure frequency.
  Proportion of patients with >50% seizure reduction in each dietary arm will be computed from daily seizure log maintained by parents
Change in social quotient with each dietary therapy | Vineland Social Maturity Scale will be done for each child at baseline and at 24 weeks to calculate social quotient at baseline and 24 weeks
  Proportion of children with improvement in social quotient at 24 weeks as compared to baseline measured by Vineland Social Maturity scale
Proportion of patients with different clinical adverse events in each group | Each child will be monitored for adverse effects clinically at 12 weeks and 24 weeks
  Each participant will be monitored clinically for adverse effects like nausea, vomiting, constipation
Correlate seizure frequency change at 24 weeks with blood HbA1c levels | Absolute level of HbA1c levels (in percentage) as compared to percentage change in seizure frequency at 3 and 6 months will be computed
  Absolute level of blood HbA1c(in percentage) as compared to percentage change in seizure frequency at 3 and 6 months will be computed
Correlate seizure frequency change at 24 weeks with blood betahydroxy butyrate levels levels | Blood beta hydroxyl butyrate levels(milimoles/liter) at 12 and 24 weeks as compared to percentage change in seizure frequency will be computed
  Blood beta hydroxyl butyrate levels(milimoles/liter) at 12 and 24 weeks as compared to percentage change in seizure frequency will be computed
Proportion of patients with different biochemical adverse events in each group | Each child will be monitored by certain biochemical investigations like hemoglobin, liver and renal function tests and lipid profile at baseline, at 24 weeks and also in between if clinically indicated
  Each participant will be monitored for side effects like anemia, dyslipidemia, deranged liver and renal function tests

CONTACTS AND LOCATIONS:
Overall Officials: Sheffali Gulati, M.D., Principal Investigator — AIIMS, New Delhi
Locations (1):
- AIIMS, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Panda PK, Chakrabarty B, Jauhari P, Sharawat IK, Agarwal A, Jain V, Pandey RM, Gulati S. Efficacy of daily versus intermittent low glycemic index therapy diet in children with drug-resistant epilepsy: A randomized controlled trial. Epilepsy Res. 2024 Mar;201:107322. doi: 10.1016/j.eplepsyres.2024.107322. Epub 2024 Feb 15. PMID 38402708